CLINICAL TRIAL: NCT02456441
Title: The Effects of Transcutaneous Tibial Nerve Stimulation in Sympathetic and Parasympathetic System in Women With Overactive Bladder: Randomized Clinical Trial
Brief Title: Effects of TENS in Autonomous System in Women With Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Luís Henrique Telles da Rosa, Clinical professor and vice-rector, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE 17136213.0.0000.5345
Record Dates: First submitted 2015-04-06; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Will be obtained the evolution parasympathetic and sympathetic system 10 minutes after TENS application, through Heart Hate Variability analysis.
  Interventions: Other: Intervention group
- Placebo group (Placebo Comparator): Will be obtained the evolution parasympathetic and sympathetic system 10 minutes after placebo current application, through Heart Hate Variability analysis. p. The placebo group will receive transcutaneous electric stimulation, for 30 seconds and then will gradually decrease by 15 seconds to not pass any current. This approach will aim to masking of the subject.
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Intervention group — The device current generator TENS used was " Neurodyn Portable Tens / Fes " of IBRAMED brand. Two self-adhesive electrodes, one immediately behind the medial malleolus and the other 10 cm above will be used. Through a chain of 1Hz, the aim is to correctly identify the tibial nerve. This position is confirmed with the rhythmic movement of the finger flexion. The frequency is then changed to 10Hz, the pulse width set at 200 "microseconds" and adjusted according to the intensity threshold for each patient, below motor threshold. This current generator also has a device, the VIF (variation in intensity and frequency) that aims to ease the accommodation of sensory receptors and enhance its effects. The application time is 30 minutes
  Other Names: Transcutaneous electric stimulation
  Arms: Intervention group
Other: Placebo group — The placebo group received an active current for 15 seconds by means of an apparatus also IBRAMED brand externally similar to that used in GI. Two self-adhesive electrodes, one immediately behind the medial malleolus and the other 10 cm above will be used.The application time for GP also was 30 minutes .
  Other Names: GP
  Arms: Placebo group

SUMMARY:
The International Continence Society (ICS) defines overactive bladder ( OAB) as a clinical syndrome characterized by urgency with or without urge incontinence , usually accompanied by frequency and nocturia , since in the absence of proven infection or other pathology related . The negative impact on quality of life of patients with OAB is already known. The etiology and pathophysiology of OAB are not completely understood. However, studies indicate an alteration of sympathetic and parasympathetic nerve stimulation involved in the mechanism of OAB. A Transcutaneous Electrical stimulation of the Tibial Nerve ( TENS) has been studied as a noninvasive and inexpensive , treating the symptoms of this syndrome therapeutic way . However, no studies in the literature evaluating the effect of electroconvulsive therapy on the mechanisms involved in sympathetic and parasympathetic modulation in these women . The objective of this study is to investigate the effects of TENS on the sympathetic and parasympathetic system in women with OAB . This is a randomized, double -blind , which will be assessed , first, in a pilot study , 30 female patients with OAB randomly allocated into 2 groups : TENS group and placebo group. Interventions take place in one day assessment of the sympathetic and parasympathetic nervous system are performed . After collecting the data will be analyzed in accordance with the statistical analysis.

DETAILED DESCRIPTION:
Hypothesis True:Electrical stimulation of the tibial nerve (TENS) decreases the activity of the parasympathetic nervous system and increases the activity of the sympathetic nervous system in women with overactive bladder.

Null Hypothesis: The electrical stimulation of the tibial nerve (TENS) does not decrease the activity of the parasympathetic nervous system and does not increase the activity of the sympathetic nervous system in women with overactive bladder.

Alternative Hypothesis: The electrical stimulation of the tibial nerve (TENS) increases the activity of the parasympathetic nervous system and decreases the activity of the sympathetic nervous system in women with overactive bladder.

Intervention Programmes

The randomization technique is carried out through sequential numbers kept in opaque envelopes, not translucent and closed. This takes into account that a major goal of randomization is to prevent the researcher to identify which intervention will be performed in each patient. The generation of sequence numbers will be made by researcher "blind" the study after patient selection criteria for inclusion and exclusion. The sequence of numbers to be used for randomization will be kept confidential until the exact moment of the beginning of the intervention.

In this study, two self-adhesive electrodes, one immediately behind the medial malleolus and the other 10 cm above will be used. Through a chain of 1Hz, the aim is to correctly identify the tibial nerve. This position is confirmed with the rhythmic movement of the finger flexion. The frequency is then changed to 10Hz, the pulse width set at 200 "microseconds" and adjusted according to the intensity threshold for each patient, below motor threshold. This current generator also has a device, the VIF (variation in intensity and frequency) that aims to ease the accommodation of sensory receptors and enhance its effects. The application time is 30 minutes.

The placebo group will receive active current for 30 seconds and then will gradually decrease by 15 seconds to not pass any current.

It is noteworthy that all study participants will be instructed not to eat, not drink, not smoke and do not exercise two hours prior to data collection.

Evaluation of the sympathetic and parasympathetic system For the analysis of Heart Rate Variability (HRV) time series of RR intervals obtained from continuous ECG signal recorded (sampling frequency = 1 kHz) for the MP150 system (Biopac, California, USA) will be interpolated and decimated to obtain equally spaced in time series and then subjected to a Fast Fourier Transform (FFT) algorithm developed using a Matlab (Matlab 6.0, Mathworks Inc., USA) language. The spectral power is calculated by integrating each frequency band of interest. The time series of RR will be analyzed in the time domain and the frequency and variability parameters and autonomic balance will be obtained. In the time domain we calculate the mean values of RR intervals, standard deviation and the square root of the sum of the square of successive differences (rMSSD). The evaluation of the sympathetic and parasympathetic nervous system will be held at the Federal University of Health Sciences of Porto Alegre (UFCSPA), the Laboratory of Physiology before, during and after application of TENS.

Calculation Sample

Due to lack of studies relating to study the effects of the sympathetic and parasympathetic TENS in women with overactive bladder nervous system, a pilot study will be conducted which will consist of:

Group A: TENS Group, composed of 15 women with overactive bladder and Group B: placebo group, consisting of 15 women with overactive bladder.

Based on the obtained values the actual sample size calculation for the study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 60 years;
* Clinical Diagnosis of Overactive Bladder Syndrome non neurogenic type;
* Score Questionnaire OAB-V8, sum equal to or greater than eight (8);
* Calendar indicating voiding more than 8 micturitions in 24 hours;
* Complaints of urinary urgency.

Exclusion Criteria:

* With a diagnosis of lower urinary tract;
* Signs of leukorrhea / diagnosis of vaginitis;
* Pregnant women;
* Diagnosed with bladder cancer and other pelvic organs;
* With a history of pelvic radiotherapy;
* With change in the sensitivity of the pelvis and lower limbs region;
* With Diabetes Mellitus;
* With known neurologic diseases;
* Patients on medications that may affect the autonomic nervous system, including anticholinergics, alpha-adrenergic antagonists, tricyclic antidepressants, serotonin, antimuscarinic, beta-receptor agonists or antagonists and antihypertensive agents;
* Use of cardiac pacemakers.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Parasympathetic and sympathetic system values obtained from heart rate variability (HRV) after TENS application | 50 minutes
  For the analysis of HRV time, series of RR intervals obtained from continuous ECG signal recorded (sampling frequency = 1 kHz) for the MP150 system (Biopac, California, USA) will be interpolated and decimated to obtain equally spaced in time series and then subjected to a Fast Fourier Transform (FFT) algorithm developed using a Matlab (Matlab 6.0, Mathworks Inc., USA) language. The spectral power is calculated by integrating each frequency band of interest. The time series of RR will be analyzed in the time domain and the frequency and variability parameters and autonomic balance will be obtained. In the time domain we calculate the mean values of RR intervals, standard deviation and the square root of the sum of the square of successive differences (rMSSD).

CONTACTS AND LOCATIONS:
Overall Officials: Luís T da Rosa, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre; Caroline HL de Lima, Msc, Study Chair — Federal University of Health Science of Porto Alegre; Patrícia V da Rosa, PhD, Study Director — Federal University of Health Science of Porto Alegre; Rodrigo DM Plentz, PhD, Study Director — Federal University of Health Science of Porto Alegre; Cinara Stein, PhD, Study Chair — Federal University of Health Science of Porto Alegre; Fabrício E Macagnan, PhD, Study Chair — Federal University of Health Science of Porto Alegre
Locations (1):
- Caroline Helena Lazzarotto de Lima, Frederico Westphalen, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Rosier PF, Hosker GL, Szabo L, Capewell A, Gajewski JB, Sand PK; International Consultation on Incontinence 2008 Committee on Dynamic Testing. Executive Summary: The International Consultation on Incontinence 2008--Committee on: "Dynamic Testing"; for urinary or fecal incontinence. Part 3: Anorectal physiology studies. Neurourol Urodyn. 2010;29(1):153-8. doi: 10.1002/nau.20762. PMID 19693957
- [Background] de Groat WC. Integrative control of the lower urinary tract: preclinical perspective. Br J Pharmacol. 2006 Feb;147 Suppl 2(Suppl 2):S25-40. doi: 10.1038/sj.bjp.0706604. PMID 16465182
- [Background] Ben-Dror I, Weissman A, Leurer MK, Eldor-Itskovitz J, Lowenstein L. Alterations of heart rate variability in women with overactive bladder syndrome. Int Urogynecol J. 2012 Aug;23(8):1081-6. doi: 10.1007/s00192-012-1738-7. Epub 2012 Apr 11. PMID 22491716
- [Background] Coyne KS, Zyczynski T, Margolis MK, Elinoff V, Roberts RG. Validation of an overactive bladder awareness tool for use in primary care settings. Adv Ther. 2005 Jul-Aug;22(4):381-94. doi: 10.1007/BF02850085. PMID 16418145
- [Background] Banakhar MA, Al-Shaiji TF, Hassouna MM. Pathophysiology of overactive bladder. Int Urogynecol J. 2012 Aug;23(8):975-82. doi: 10.1007/s00192-012-1682-6. Epub 2012 Feb 7. PMID 22310925
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Fall M, Lindstrom S. Electrical stimulation. A physiologic approach to the treatment of urinary incontinence. Urol Clin North Am. 1991 May;18(2):393-407. PMID 2017820